CLINICAL TRIAL: NCT05199519
Title: A Phase Ia Study to Evaluate the Safety, Tolerance, Pharmacokinetics and Preliminary Efficacy of IBI345 in Patients With CLDN18.2-positive Solid Tumors
Brief Title: Study to Evaluate the Safety, Tolerance, Pharmacokinetics and Preliminary Efficacy of IBI345
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI345Y001
Record Dates: First submitted 2021-11-28; First posted 2022-01-20 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: CLDN18.2 Positive Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBI345 (Other): Single arm
  Interventions: Drug: IBI345

INTERVENTIONS:
Drug: IBI345 — IBI345 CAR-T cell injection by intravenous infusion

SUMMARY:
A phase Ia study to evaluate the safety, tolerance, pharmacokinetics and preliminary efficacy of IBI345 in patients with CLDN18.2 positive solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤75 years.
2. Histologically or cytologically confirmed CLDN18.2 positive patients with advanced gastric cancer or pancreatic cancer who failed standard therapy .
3. There are assessable lesions according to RECIST V1.1 (solid tumor efficacy evaluation criteria).
4. Expected survival time ≥12 weeks.
5. ECOG PS 0~1.

Exclusion Criteria:

1. Participating in another interventional clinical study, other than observational (non-interventional) clinical study or in the survival follow-up phase of the interventional study.
2. Received any antitumor drug within 2 weeks prior to apheresis or initial administration of the investigational drug.
3. Use of immunosuppressive drugs within 1 week prior to apheresis or 2 weeks prior to initial administration of the investigational drug.
4. Long-term systemic steroid or any other immunosuppressive drug therapy is required, not including inhaled steroid therapy.
5. Receive live attenuated vaccine within 4 weeks prior to initial administration of the study drug or plan to receive live attenuated vaccine during the study period.
6. Toxicity (excluding alopecia, fatigue, and hematological toxicity) that did not return to equal to or lower than Grade 1 of NCI CTCAE V5.0 from previous antitumor therapy prior to initial administration of the investigational drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-10-29 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | up to 2 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) according to RECIST version 1.1 | up to 2 years
  Defined as the proportion of subjects with confirmed complete response (CR) or partial response (PR); a confirmed response is a response that persists on repeat-imaging ≥4 weeks after initial documentation of response.
Duration of Response (DOR) according to RECIST version 1.1 | up to 2 years
  Defined as time from date of first objective response (either CR or PR) to first documentation of radiographic disease progression or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) according to RECIST version 1.1 | up to 2 years
  Defined as the proportion of subjects who have achieved CR, PR, or stable disease (duration of stable disease should be ≥3 months).
Time to Response (TTR) according to RECIST version 1.1 | up to 2 years
  Defined as the time from first dose to first documentation of objective response (either CR or PR).
Progression-Free Survival (PFS) according to RECIST version 1.1 | up to 2 years
  Defined as the time from first dose to first documentation of radiographic disease progression or death due to any cause, whichever occurs first.
Overall Survival (OS) according to RECIST version 1.1 | up to 2 years
  Defined as the time from first dose to the date of death due to any cause.
Peak Plasma Concentration (Cmax) | up to 1 years
Area under theplasma concentration versus time curve (AUC) | up to 1 years
Time of maximum drug concentration in hours [Tmax] | up to 1 years
Elimination half-life in hours [t1/2] | up to 1 years
Clearance (CL) | up to 1 years
Distribution Volume (Vd) | up to 1 years
Number of Participants With anti-drug antibody (ADA) | up to 1 years
Number of Participants With Neutralizing Antibodies (NAbs) | up to 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No